CLINICAL TRIAL: NCT06812702
Title: A Multi-site Longitudinal Cohort Study of Prodromal and Clinical Parkinson'sDisease
Brief Title: Parkinson's Disease Biomarker Study
Acronym: PDBS
Status: Recruiting | Type: Observational
Sponsor: Ronald Postuma (Other)
Responsible Party: Sponsor-Investigator, Ronald Postuma, MD, MSc, McGill University
Organization: McGill University (Other)
Other Study IDs: PDBS
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease, Idiopathic; REM Sleep Behavior Disorder
MeSH Terms: conditions — Parkinson Disease; REM Sleep Behavior Disorder | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Optional skin biopsy will be collected paravertebrally at approximately the C8 level at baseline. This procedure is performed to validate an immunohistochemistry skin biopsy assay for the detection of pathological alpha-synuclein diagnostic of PD. Follow up skin samples of consenting participants will be collected at the one-year follow-up.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Control: Above 40 years of age, sex matched with PD cohort. Participants may consent to additional skin biopsy at baseline and at the one-year follow-up. Skin will be taken paravertebrally at approximately the C8 level.
  Interventions: Other: Observational; Procedure: Skin Biopsy
- RBD Patients: Polysomnographic confirmed RBD, age 50 years or older, male and female. RBD patients only will receive DaT-SPECT and MRI imaging at baseline and Week52 of the study. Participants may consent to additional skin biopsy at baseline and at the one-year follow-up. Skin will be taken paravertebrally at approximately the C8 level.
  Interventions: Other: Observational; Procedure: Skin Biopsy
- PD patients: Patients with PD first diagnosed 2-6 years prior to enrolment, above 40 years of age, male and female. Participants may consent to additional skin biopsy at baseline and at the one-year follow-up. Skin will be taken paravertebrally at approximately the C8 level.
  Interventions: Other: Observational; Procedure: Skin Biopsy

INTERVENTIONS:
Other: Observational — Observational
Procedure: Skin Biopsy — Participants may consent to additional skin biopsy at baseline and at the one-year follow-up. Skin will be taken paravertebrally at approximately the C8 level.

SUMMARY:
The primary objective of this study is to determine whether data acquired from a remote monitoring approach can reliably identify and track motor symptoms in prodromal PD and clinical PD.

The study is a one-year longitudinal biomarker study recruiting idiopathic RBD patients, Parkinson's Disease patient and healthy controls. All participants receive a smartphone with the Roche PD Mobile Application, complete a number of active tests daily and their movements will be remotely monitored. Participants will undergo additional neurological exams and DaT-SPECT and MRI imaging in the study.

A second objective of this study will be to validate an immunohistochemistry skin biopsy assay for the detection of pathological alpha-synuclein diagnostic of PD, in the peripheral nerves of the skin.

ELIGIBILITY:
Inclusion Criteria:

* signed consent form, male or female over age 40, ability to follow protocol, additional group-specific inclusion criteria

Exclusion Criteria:

* participation in interventional clinical study within 3 months of screening, moderate to severe depression in judgement of the investigator, any concomitant disease, condition or treatment which may interfer with the conduct of study (determined by investigator), additional group-specific exclusion criteria

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: male or female over age 40, ability to follow protocol
Sampling Method: Non-Probability Sample
Enrollment: 295 (Estimated)
Dates: Start 2019-03-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Digital Biomarkers | 12 months
  Changes in continuous sensor-based measurements derived from Roche PD MobileApplication, with active testing and passive monitoring in idiopathic RBD and clinical PD (1 month in Healthy Controls)

SECONDARY OUTCOMES:
alpha-synuclein deposition in skin biopsy | 12 months
  Frequency of pathological alpha-synuclein deposition in the skin biopsy assay in idiopathic RBD and clinical PD and HC (optional study procedure)
Changes in sensor-based measurements and passive monitoring | 12 months
  Relationship between changes in continuous sensor-based measurements derived from Roche PD Mobile Application active testing and passive monitoring over 12 months in idiopathic RBD, clinical PD and HC and changes in clinical assessments
Correlation of sensor-based measurements and imaging outcomes | 12 months
  For idiopathic RBD patients only, correlation between sensor-based measurements derived from Roche PD Mobile Application active testing and passive monitoring and changes in MRI and DaT-SPECT outcome measures.

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - Pacific Parkinson's Research Centre, Vancouver, British Columbia
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - The Neuro, Montreal, Quebec
  - Centre de recherche du CHU de Québec-Université Laval (CHUQ), Québec

IPD SHARING:
Plan to Share IPD: No